CLINICAL TRIAL: NCT00959556
Title: Search for Genetic Factors Predictive of Response to Chemotherapy in Patients With or Who Has a Mammary Adenocarcinoma in Neo-adjuvant or Metastatic Setting
Brief Title: Study of Blood Samples in Patients With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000633531; COL-GENEOM; COL-IDRCB-2007-A00908-45; COL-2007-08; INCA-RECF0635
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying the genes expressed in samples of blood from patients with cancer may help doctors identify biomarkers related to cancer. It may also help doctors predict how patients will respond to chemotherapy.

PURPOSE: This clinical trial is studying blood samples in patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify constitutional gene variants associated with a change in response.

OUTLINE: Blood samples are collected periodically for analysis of genetic factors.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast carcinoma
* Received first-line chemotherapy (in neoadjuvant or metastatic setting) comprising anthracyclines and/or taxanes, including for a second primary cancer
* Patient agrees to conservative surgery
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* No contraindication for chemotherapy comprising anthracyclines and/or taxanes

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior adjuvant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Histologic complete response (Chevallier and Sataloff) or tumor response (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Bonneterre, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France